CLINICAL TRIAL: NCT04288700
Title: Evaluation of the Efficacy of Captopril Versus Propranolol and Timolol as a Treatment of Infantile Capillary Hemangioma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Mohamed El-Sayed Ibrahim Atta, Teaching Assistant, Pharmacy Practice and Clinical Pharmacy Department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 257
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Infantile Hemangioma
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Propranolol; Captopril; Timolol; Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator)
  Interventions: Drug: oral propranolol
- Group B (Active Comparator)
  Interventions: Drug: Oral Captopril
- Group C (Active Comparator)
  Interventions: Drug: intralesional propranolol injection
- Group D (Active Comparator)
  Interventions: Drug: topical Timolol maleate 0.5% eye drops

INTERVENTIONS:
Drug: oral propranolol — oral propranolol therapy at a dose of 1 mg/kg/d (Inderal 20 mg/5 mL) in three divided doses. If the child will tolerate the treatment with no side effects, therapy will continue in an outpatient clinic. Blood glucose level will be also measured in a periodic manner during therapy. The dose will be increased gradually to 2 mg/kg/d in three divided doses if there will be no adverse effects from the initial therapy.
  Arms: Group A
Drug: Oral Captopril — A test dose of 0.1 mg kg) will be administered orally with pulse rate and blood pressure monitored at 0.5, 1 and 2 h and at each follow up. If the test dose is tolerated, captopril administration will start at 0.15 mg kg) per dose 8-hourly. Pulse rate and blood pressure will be monitored 4-hourly and doses will be withheld if hypotension is documented. After 24 h, the dose will be increased to 0.3 mg kg) per dose 8-hourly .
  Arms: Group B
Drug: intralesional propranolol injection — intralesional propranolol injection 1 mg/mL
  Arms: Group C
Drug: topical Timolol maleate 0.5% eye drops — To be Applied on the surface of the lesions three times daily
  Arms: Group D

SUMMARY:
Is to compare and evaluate the efficacy of oral captopril with oral propranolol, intralesional propranolol injection, and topical Timolol in the treatment of infantile hemangioma and their effect on vascular endothelial growth factor and CD 133.

DETAILED DESCRIPTION:
Infantile hemangiomas are the most common benign tumor of infancy, affecting up to 10% of the pediatric population with a higher incidence in female (3:1), preterm infants, and Caucasian population. The molecular mechanisms underlying pathogenesis remain incompletely understood, but the clinical course follows a stereotyped pattern: a phase of early vascular proliferation over the first year of life followed by a gradual phase (1 to7 years in duration) of spontaneous involution and replacement of vascular channels by fibro-fatty tissue. Despite their benign nature,in certain cases IHs can cause severe morbidities and therefore sometimes require medical intervention.

Vascular endothelial growth factor A is the predominant growth factor associated with endothelial proliferation, migration, and survival. Vascular endothelial growth factor, being a potent inducer of vascular permeability, is known to cause edema and lead to formation of hemangiomas in high concentrations along with CD133 is a transmembrane glycoprotein which represents a cell surface marker for hemangioma-derived stem cells (HemSCs). CD133-positive HemSCs can still be diﬀerentiated into hemangiomas, suggesting that CD133-positive HemSCs have continuous ability to form hemangiomas. Targeted elimination of CD133-positive HemSCs could fundamentally inhibit the proliferation of hemangioma.

Aim of the study is to compare and evaluate the efficacy of oral captopril with oral propranolol, intralesional propranolol injection, and topical Timolol in the treatment of infantile hemangioma and their effect on vascular endothelial growth factor and CD 133.

Methodology : Open label Randomized Controlled trail will be carried out at Vascular malformation clinic of Pediatric Surgery department of Ain Shams University ,Patients of the study will be randomly allocated equally into 4 groups (A, B, C, D), 25 patients each.

* Group A: Subjected to oral propranolol therapy at a dose of 2 mg/kg/d in three divided doses.
* Group B: Oral Captopril will be administered as a test dose of 0.1 mg kg orally with pulse rate and blood pressure monitored at 0.5, 1 and 2 h and at each follow up. If the test dose is tolerated, captopril administration will start at 0.15 mg/ kg) per dose 8-hourly. Pulse rate and blood pressure will be monitored 4-hourly and doses will be withheld if hypotension is documented. After 24 h, the dose will be increased to 0.3 mg/ kg) per dose 8-hourly.
* Group C: Subjected to intralesional propranolol injection 1 mg/mL. The volume of injected drug depends on the size of the lesion (0.2 mL will be injected per cm of lesion diameter), with a maximum volume of 1 mL for a lesion of 5 cm diameter
* Group D: Subjected to topical Timolol maleate 0.5% eye drops on the surface of the lesions three times daily and gentamycin ointment will be applied around the lesions to prevent the timolol from leaking.

Following up: Venous blood samples will be withdrawn from all study participants at study entry and after 6 months of treatment for assessment of serum levels of VEGF and CD 133 by ELISA technique along with the size of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients younger than 12 years and older than 2 months of age with infantile hemangioma

Exclusion Criteria:

* Patient with ulcerated or infected hemangioma.
* Patient younger than 2 months and older than 12 years of age.
* Patients with multiple hemangiomas.
* Any Patient with cardiovascular problems, bronchial asthma, diabetes mellitus, bilateral renal stenosis, Electrolyte disturbance, or renal impairment was excluded.
* Patients with abnormal electrocardiogram, or echocardiogram should be excluded.
* Patients who have had previous treatment for hemangioma.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of serum levels of Vascular endothelial growth factor | 6 months
Assessment of serum levels of CD 133 | 6 months
Assessment of the size of the lesion. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rana Atta, BSc, Principal Investigator — Future University in Egypt
Locations (1):
- Vascular malformation clinic of Pediatric Surgery department of Ain Shams University., Cairo, Egypt